CLINICAL TRIAL: NCT03373032
Title: Skin Sensitivity Acupuncture and Kinesiotherapy on Breast Cancer Patients Subject to Chemotherapy With Taxans
Acronym: Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Gil Facina, Professor Doctor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FUSaoPaulo,PT 6
Record Dates: First submitted 2017-11-09; First posted 2017-12-14 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Chemotherapy Effect
Keywords: Physical Activity; Sensory Neuropathy; Acupuncture; Depression; Anxiety; Skin Sensitivity
MeSH Terms: conditions — Motor Activity; Depression; Anxiety Disorders | interventions — Acupuncture Therapy; Exercise; Observation

STUDY DESIGN:
Intervention Model Description: A computer program will produce a randomization list, which will generate random sequences for the three groups and will be recorded and placed in sealed, opaque, non-translucent and sequentially numbered envelopes. This intervention should be done by someone else and not by the principal investigator. These envelopes will be opened after the consent of the patient to participate in the research and only then will the researcher know as well as the patient the group that she will be allocated. 124 envelopes were available where 31 would contain code that allocates the patients in group A, 31 in group B, 31 in group C or 31 group Follow Up .No Intervention Group - S 'Class wait '. This was done in order to avoid influences such as the therapist's or patient's preferences related to the intervention.
Who Masked: Participant
Masking Description: Blind ramdomization and blind final evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Stiper - A (Experimental): Stiper, breast cancer patients during chemotherapy cycles, once a week, during 10 weeks
  Interventions: Other: Stiper
- Acupuncture - B (Experimental): Acupuncture with needles, breast cancer patients during chemotherapy cycles, once a week, during 10 weeks
  Interventions: Other: Acupuncture
- Exercise - C (Experimental): Exercise, breast cancer patients during chemotherapy cycles, once a week, during 10 weeks
  Interventions: Other: Exercise
- Follow Up - D (Experimental): Selected patients from the 3 groups Stiper / Acupuncture / Exercise. One session with a Peridell Massager
  Interventions: Other: Follow Up
- Observation - S (Other): Group patients who were unable to participate in the intervention group A / B and C. In this group, only the evaluation will be performed.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Stiper — Stiper silicon tablets, for acupunture's stimulation of meridian points, the Stiper's chemical composition is nothing more than SiO 2 - (silicon dioxide) the shape of the quartz stone (silicon rich).They will perform the treatment with the "Stiper" silicon inserts, which will be applied and fixed by plasters at the acupuncture points, duration of 05 minutes.
  Arms: Stiper - A
Other: Acupuncture — Treatment with a systemic needle to stimulate meridian acupuncture points, treatment begins with asepsis with 70% alcohol-soaked cotton in the region of the acupoints and then sterile and disposable needles (0.25 mm x 30 mm) will be inserted in both limbs, will be placed in the following regions: shoulders, thorax, legs and feet with the puncture order from bottom to top,duration of 30 minutes.
  Arms: Acupuncture - B
Other: Exercise — Will perform pre-defined kinesiotherapy based on the stretching of cervical musculature and scapular waist, lumbar spine and lower limbs with exercises for WM and upper limb (MS) and lower limb (MI) strength with a duration of 30 minutes.
  Arms: Exercise - C
Other: Follow Up — Use of the therapeutic massager, in hands and feet, to stimulate region's sensitivity, women who were submitted to the chemotherapy treatment with Taxane and continued with changes in sensitivity. Once in each dermatome, adding time of 5 minutes of application on average.
  Arms: Follow Up - D
Other: Observation — The waiting room (observation) group did not receive any intervention. Conduct evaluations of the research protocol as groups A, B and C.
  Other Names: Control
  Arms: Observation - S

SUMMARY:
Objective: to compare different therapies employing acupuncture needles, silicon pellets and kinesiotherapy in breast cancer patients to taxane chemotherapy cycles. Methods:The present study will be carried out at the Oncomastology outpatient clinic of the UNIFESP (Federal University of São Paulo) Gynecology Department's Discipline of Mastology - Escola Paulista de Medicina (EPM) and the Oncology Clinic Associated Center of Oncology, located at Rua Gabriel Monteiro da Silva, 454. randomized clinical trial will be conducted to define the treatment. Patients will be allocated into three groups (Group A: Stiper, Group B: Acupuncture, Group C: Kinesiotherapy and Group D After treatment ) who will receive treatment once a week for eight consecutive weeks. Group - S-observation.124 patients will be randomized in one of the three groups, after having signed the Free and Informed Consent Form and agreed to participate in the project, will respond to the evaluation form and will be submitted to physical examination. Patients will be evaluated in the first and tenth sessions.

Keywords: Acupuncture, Breast Neoplasm, Chemotherapy.

DETAILED DESCRIPTION:
Women will be recruited at the Oncomastology outpatient clinic of the UNIFESP (Federal University of São Paulo) Gynecology Department's Discipline of Mastology - Escola Paulista de Medicina (EPM) and Clínica de Oncologistas Associados Centro Integrado de Oncologia, located at Rua Gabriel Monteiro da Silva, 454. Patients will consecutively be selected by order of entry in the chemotherapy recorded in the log and randomized in one of three intervention groups. Complying with all the research's ethical aspects, the following procedures will apply: 1st clarify the study's objectives;2nd sign the Term of Free and Informed Consent, signed in two ways, as one stays with the patient; 3rd espond to the evaluation form in the following items: socioeconomic aspects, main complaint, family history, personal history, surgical data, pathological anatomy, radiotherapy, chemotherapy, hormone therapy, sensitivity and perimetry;4 th physical exams. Completed the FACT-TAXANE questionnaire. Patients will be evaluated in the first and tenth sessions.

ELIGIBILITY:
Inclusion Criteria:

* women over 18 years old
* women submitted to chemotherapy with taxanes
* the 1th cycle both neoadjuvant and adjuvant with staging from I to III no mental changes

Exclusion Criteria:

* Women with preexisting diseases such as locoregional or distant cancer, previous joint pain,
* rheumatic disease,
* who are not undergoing chemotherapy with Anthracyclics and / or Cisplatin
* acupuncture in another service in the last three will be excluded.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female breast cancer patients under taxanes based chemotherapy
Enrollment: 79 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Measure sensitivity changes | One day, Two weeks, Ten weeks
  It will be evaluated with an estiometer for sensitivity changes (green, blue, violet, red, orange, pink) the lighter color green represents a better sensitivity and as this color becomes darker it represents a worsening of sensitivity reaching the pink color.
  Visual Scale 0-10 0 no pain and 10 unbearable pain
Tongue inspection Changes | Baseline, Ten Weeks
  Tongue assessments will be recorded by photograph before and after treatment and the following characteristics will be observed: Humidity, Color, Coating, Size, Movement, Other findings.

SECONDARY OUTCOMES:
Questionnaires FACT G + TAXANES | Baseline, Ten Weeks
  To derive a FACT-Taxane Trial Outcome Index (TOI) Score range: 0-120 To Derive a FACT-G total score Score range: 0-108 To Derive a FACT-Taxane total score Score range: 0-172
Sensitivity changes with peridell | One day
  Intervention session using a massager Peridell®️ therapy, with subsequent reassessment of sensitivity.
Pain MC Gill | Baseline, Ten Weeks
  These four groups are organized into 20 subgroups according to the painful sensation. Subgroups 1 to 10 represent sensitive responses to the painful experience (traction, heat, torsion, among others): the descriptors of subgroups 11 to 15 are affective responses (fear, punishment, neurovegetative responses, etc.). Subgroup 16 is evaluative (assessment of the overall experience) and those from 17 to 20 are miscellaneous.
Beck Depression Inventory (BDI) | Baseline, Ten Weeks
  The higher the total score of the Inventory, the worse the depressive state of the patient. This score is classified according to 4 bands that define the degree of patient's depression (from 0 to 13: No Depression; from 14 to 19: Mild Depression; from 20 to 28: Moderate depression; 29 to 63: Severe Depression).

OTHER OUTCOMES:
Beck Anxiety Inventory (BAI) | Baseline, Ten Weeks
  The score is classified according to 4 ranges that define the patient's degree of anxiety (from 0 to 7: Minimum Anxiety; from 8 to 15: Mild Anxiety; from 16 to 25: Moderate Anxiety; 26 to 63:
  Severe Anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Gil Facina, PHD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Brazil Federal University São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No